CLINICAL TRIAL: NCT02458820
Title: Prompt Diagnosis and Treatment of Subclinical Seizures After Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-011635; 5K23NS075363 (NIH)
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Heart Arrest; Seizures
Keywords: Cardiopulmonary Resuscitation; Return of Spontaneous Circulation; ROSC; Electroencephalogram
MeSH Terms: conditions — Heart Arrest; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Patients will be recorded and interpreted as per standard of care. If a seizure is noted by the neurology service, the standard seizure treatment protocol will be used by the clinical team.
- DSA EEG + Usual Care (Experimental): Patients will undergo at least hourly interpretation of DSA by the ICU bedside care provider. If the bedside care provider is concerned that there is a seizure on DSA they will contact the EEG tech on call for confirmation. If a seizure is confirmed by neurology, the standard seizure treatment protocol will be used by the clinical team.
  Interventions: Procedure: DSA EEG

INTERVENTIONS:
Procedure: DSA EEG — Color density spectral array (DSA) is a quantitative electroencephalogram (EEG) technique that uses Fourier transformation to present EEG power (amplitude2/Hz, by color) and frequency (y-axis) over time (x-axis). It is commercially available and used routinely by neurophysiologists for EEG interpretation. Up to several hours of EEG can be displayed as a single image.
  Other Names: Color density spectral array electroencephalogram
  Arms: DSA EEG + Usual Care

SUMMARY:
Non-convulsive seizures (NCS) following cardiac arrest are common and are associated with worse neurologic outcomes and increased mortality. More prolonged seizures (status epilepticus) are associated with worse outcomes. Earlier diagnosis and treatment of seizures may lead to earlier termination of seizures and decreased seizure burden.

This study will evaluate whether bedside intensive care unit (ICU) provider interpretation of a type of EEG called DSA EEG can be used by non-neurologists to diagnosis seizures more rapidly than continuous EEG's routinely read by neurologists.

DETAILED DESCRIPTION:
Acute symptomatic electroencephalographic (EEG) seizures are common in children who experience a cardiac arrest, and are associated with worse short term survival. In larger studies of critically ill children with heterogeneous acute encephalopathy etiologies, EEG seizures occur in 10-40% of monitored patients, and there is increasing evidence that high seizure burdens are associated with worse outcomes. Furthermore, status epilepticus treatment delays are associated with reduced medication efficacy for status epilepticus termination. The majority of EEG seizures in critically ill children have no clinical correlate and therefore detection requires EEG monitoring. Many institutions do not have access to continuous EEG monitoring services. Additionally, even when EEG "monitoring" is performed, data review is generally intermittent, leading to delays between seizure onset and detection.The purpose of the study is to determine the efficacy of real-time DSA pattern interpretation for the detection of seizures by bedside ICU practitioners.The primary objective of this study is to determine the whether the real-time DSA patterns interpreted by bedside ICU practitioners can decrease the time to accurate NCS detection following pediatric cardiac arrest. All subjects who receive chest compressions and have return of spontaneous circulation and are cared for the CHOP Pediatric Intensive Care Unit (PICU) will be screened. If patients meet inclusion criteria they will be approached for consent. Written informed consent will be obtained from parents/guardians. Assent will not be obtained as these children are intubated and comatose after arrest.Patients will be randomly assigned to receive standard of care, continuous EEG monitoring, versus continuous EEG monitoring plus real-time ICU provider DSA interpretation. This will go on for the duration of clinically indicated EEG monitoring.

For patients enrolled in the standard continuous EEG arm of the study, EEG will be recorded and interpreted as per standard of care. If a seizure is noted by the neurology service, the standard seizure treatment protocol will be used by the clinical team.Patients monitored with standard EEG and DSA will undergo at least hourly interpretation of DSA by the ICU bedside care provider. If the bedside care provider is concerned that there is a seizure on DSA they will contact the EEG tech on call for confirmation. If a seizure is confirmed by neurology, the standard seizure treatment protocol will be used by the clinical team.Following completion of EEG intervention arms, the patients will be followed and discharge survival and discharge Pediatric Cerebral Performance Category (PCPC) will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age > 48 hours
2. Return of Spontaneous Circulation (ROSC) for > 20 minutes after a cardiac arrest
3. Treated in the PICU
4. Clinical team ordering continuous EEG monitoring

Exclusion Criteria:

1. Age < 48 hours old and < 38 weeks gestational age
2. No available computers with DSA software

Min Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Average time from EEG seizure onset to seizure recognition | 3 days
  EEG monitoring and DSA interpretation by ICU practitioners will continue for the duration of clinically indicated EEG monitoring which will be no more than 3 days. The average time from seizure onset to seizure recognition between the EEG group and the EEG + DSA group will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Topjian, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States